CLINICAL TRIAL: NCT06260436
Title: Questionnaire About The Incidence of Lower Urinary Tract Symptoms Among a Sample of Women Before and After Surgical Correction of Uterine Prolapse and Impact on Quality of Life
Brief Title: Questionnaire of Lower Urinary Tract Symptoms Among Women Before and After Surgical Correction of Uterine Prolapse
Status: Recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Tharwat Gamal Mohammed Ibrahim, principal investigator, Assiut University
Other Study IDs: Tharwat gamal Mohamed
Record Dates: First submitted 2024-02-07; First posted 2024-02-15 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- pelvic organ prolapse patients with lower urinary tract symptoms: this group for patient who have pelvic organ prolapse and lower urinary tract symptoms
- pelvic organ prolapse patients without lower urinary tract symptoms: this group for patient who have pelvic organ prolapse but do not have any lower urinary tract symptoms

SUMMARY:
. The study will include patients who underwent Pelvic reconstructive surgery for advanced pelvic organ prolapse (POP-Q ≥ 3). Data regarding preoperative evaluation, surgical procedure, and post-operative management will be collected. women will receive a follow up questionnaire. . The baseline questionnaire included data on age, urinary incontinence, daytime frequency, nocturia, postmicturition dribble, straining, urgency, incomplete bladder emptying, and hesitancy. Women were asked about leakage caused by coughing or sneezing, moving, lifting, sleeping, sexual intercourse, urgency, and rest.

DETAILED DESCRIPTION:
Pelvic organs prolapse (POP) is defined as the downward descent of the pelvic organs resulting in protrusion of the vagina and/or uterine cervix. POP and overactive bladder (OAB) often co-exist. The International Continence Society defines OAB as "urgency with or without urge incontinence, usually with frequency and nocturia" Of women with symptomatic pelvic organ prolapse, 13-39% experience voiding dysfunction (VD).

The aim of the study is to determine the effect of prolapse surgery on voiding function. The study will include patients who underwent Pelvic reconstructive surgery for advanced pelvic organ prolapse (POP-Q ≥ 3). Data regarding preoperative evaluation, surgical procedure, and post-operative management will be collected. women will receive a follow up questionnaire.

Non-responders will send a reminder after three weeks and if the non-responders still failed to respond were eventually asked to complete a short form comprising questions on urgency and incontinence. This procedure followed guidelines outlined by the local ethical committee. The baseline questionnaire included data on age, urinary incontinence, daytime frequency, nocturia, postmicturition dribble, straining, urgency, incomplete bladder emptying, and hesitancy. Women were asked about leakage caused by coughing or sneezing, moving, lifting, sleeping, sexual intercourse, urgency, and rest. stress incontinence according to the International Continence Society defined as leakage caused by exertion (coughing or sneezing, moving, or lifting) and urge incontinence as leakage associated with urgency.

ELIGIBILITY:
Inclusion Criteria:

1. Age; greater than or equal to 18 years
2. women with urogenital prolapse grade 3 or more
3. indicated for surgical repair for pelvic organ prolapse
4. Willing and able to sign an informed consent
5. Willing to comply with the study protocol

Exclusion Criteria:

1. Anti-incontinence surgery
2. Lower urinary tract anomaly
3. Active urinary tract infections
4. Bladder tumor.
5. Bladder stones

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — only female cases will be eligible to participate
Study Population: female cases at women health hospital at assuit university
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2021-05-30 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
effect of surgical correction of pelvic organ prolapse on the lower urinary tract symptoms | 3 months
  the effect of surgical correction of pelvic organ prolapse on the lower urinary tract symptoms will be checked through a validated questionnaire before and after surgical correction

SECONDARY OUTCOMES:
effect of surgical correction of pelvic organ prolapse on the quality of life | 3 months
  the questionnaire will check the effect of surgical correction of pelvic organ prolapse on quality of life

CONTACTS AND LOCATIONS:
Overall Officials: tharwat gm mohamed, Principal Investigator — Assiut University; Mustafa mb bahlool, professor, Study Director — Assiut University
Locations (1):
- Assuit University, Asyut, Assuit, Egypt

IPD SHARING:
Plan to Share IPD: No
no data can be shared

REFERENCES:
- [Result] Baessler K, O'Neill SM, Maher CF, Battistutta D. Australian pelvic floor questionnaire: a validated interviewer-administered pelvic floor questionnaire for routine clinic and research. Int Urogynecol J Pelvic Floor Dysfunct. 2009 Feb;20(2):149-58. doi: 10.1007/s00192-008-0742-4. Epub 2008 Oct 29. PMID 18958382